CLINICAL TRIAL: NCT02209558
Title: The Effect of Visual Sternal Precautions on Behavioral Intentions and Readmissions
Acronym: Sternal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: North Shore University Hospital (Other)
Responsible Party: Principal Investigator, Craig Feinman, Senior Cardiothoraic Physical Therapist, Physical Therapy, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-305B
Record Dates: First submitted 2014-08-01; First posted 2014-08-06 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Intention - Mental Process; Readmission Rates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Written Sternal Precautions (No Intervention): Patients will receive education that is the "standard of care" at North Shore Long Island Jewish Health Systems in their post-operative sternal precautions.
- Visual Sternal Precautions (Experimental): Patients will receive both "standard of care" written sternal precautions, as well as visual sternal precautions.
  Interventions: Behavioral: Visual Sternal Precautions

INTERVENTIONS:
Behavioral: Visual Sternal Precautions — Visual depiction of SPs in addition to "standard of care" written precautions
  Arms: Visual Sternal Precautions

SUMMARY:
Sternal precautions are standard patient education protocol disseminated to post-operative open heart surgery patients . While this "best practice" safety measure is widely distributed to patients, the origin of said precautions is unknown. Statewide hospitals vary on their parameters for sternal precautions using a myriad of restrictions, i.e. weighted activities, biomechanical movements to be avoided. In addition, the medium in which sternal precautions are taught varies, thus complicating patient adherence to these vital post-operative measures.

The primary objective of this study is to use a randomized pre-post test design to compare two different training procedures. One training group examines current standard of care (providing verbal instruction using teach back and written sternal precautions). The second training group provides subjects with visual depiction of sternal precautions, in addition to standard of care. The study will analyze 30 and 60 day readmission rates for aforementioned patients. Finally, the study will assess changes in behavior intentions from before training to after training in both groups via behavioral analysis survey consisting of 8 questions.

Hypothesis 1: The investigators hypothesize that subjects provided with visual sternal precautions, in addition to standard of care, will have a lower 30 and 60 day readmission rate when compared to subjects in the standard of care group

Hypothesis 2: The investigators hypothesize that changes in behavior intentions toward sternal precautions will be greater from before training to after training in the visual SPs in addition to standard of care group than the standard of care only group.

DETAILED DESCRIPTION:
Eligible subjects will be identified by the Senior Cardiothoracic Physical Therapist (Dr. Craig D. Feinman, PT, DPT) on staff at North Shore University Hospital. Dr. Feinman will provide basic study information to potential subjects and refer those that are interested in the study to the research team who will then provide a copy of the consent form and more information about the study. Inclusion Criteria represents post-surgical adult patients who had a median or midline sternotomy incision during cardiac surgery at North-Shore University Hospital. Exclusion Criteria represents patients with dementia or those that are cognitively impaired will be excluded from the study.

A T-test or Mann Whitney U test will be use to compare group differences on continuous variables, e.g. age. Beta regression or logistic regression model will be developed for the outcomes of adherence and readmission proportions/rates. To assess changes from pre to post training on behavioral intentions a paired t-test or Wilcoxon signed rank for matched pairs will be used. A result will be considered statistically significant at the p<0.05 level of significance. All analyses will be performed using SAS version 9.3 (SAS Institute, Cary, NC).

ELIGIBILITY:
Inclusion Criteria:

* Post-surgical adult patients who had a median or midline sternotomy incision during cardiac surgery at North-Shore University Hospital.

Exclusion Criteria:

* Patients with dementia or those that are cognitively impaired will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Patient behavioral intentions post visual training strategies | Post-operative day one when patient medically cleared for PT evaluation, 2nd session, and prior to discharge from hospital (approximately 1-10 days)
  The intervention group will receive "standard of care" sternal precautions delivered via written medium. In addition, printed visual depictions of sternal precautions will be provided. During completion of the initial Physical Therapy evaluation, patients will be asked to provide baseline knowledge of sternal precautions via "teach back," an important tool in assessing patients' knowledge of important points delivered during clinical practice. Patients will then perform teach back of sternal precautions upon second Physical Therapy encounter to ensure understanding and post-operative anesthesia effects have waned. Prior to discharge (when patient deemed medically appropriate by the medical/surgical team), the patient will receive a survey consisting of 8 behavioral intention questions with "yes," "no," or "not sure" responses. Questions posed on the surveys assess if patients will/will not perform certain behaviors that may/may not predispose a risk to the patient's sternum.

SECONDARY OUTCOMES:
30 and 60 day readmission rates | 30-60 days post patient discharge from hospital setting
  Re-admission rates of enrolled subjects is integral in determining if patients adhere to sternal precautions after discharge. Resumption of regular activities is cleared by the medical/surgical team. The study team will review the medical records of the subjects 60 days after enrollment to determine if and why they were re-admitted to the hospital. Since there is a possibility for subjects to be re-admitted to facilities outside of the health system, the study team will also call the enrolled subjects 60 days after enrollment to obtain this information.

CONTACTS AND LOCATIONS:
Overall Officials: Craig D Feinman, Doctor of Physical Therapy, Principal Investigator — North Shore University Hospital, NSLIJ Health System; Renee Pekmezaris, PhD, Study Director — North Shore University Hospital, NSLIJ Health System; Andrzej Kozikowski, PhD, Study Director — North Shore University Hospital, NSLIJ Health System; Jonathan Dropkin, ScD, PT, Study Director — North Shore University Hospital, NSLIJ Health System; Joanna Steinn, MPH, Study Director — North Shore University Hospital, NSLIJ Health System; Alan Hartman, MD, Study Director — North Shore University Hospital, NSLIJ Health System
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States